CLINICAL TRIAL: NCT07030933
Title: Amino Acid Infusion in Cardiac Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Adam Adenwala, Assistant Professor of Anesthesiology, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study01
Record Dates: First submitted 2025-06-03; First posted 2025-06-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Implementation - Standard of Care (No Intervention): Participants in this group will receive their anesthetic care that is the current standard of care at our institution for patients undergoing cardiac surgery with cardiopulmonary bypass.
- Post-Implementation - Amino Acid Treatment (Experimental): Participants in this group will receive the standard of anesthetic care at our institution plus treatment of amino acid infusion (Travesol 10%, Baxter) at a dose of 2g per kilogram of ideal body weight per day until their discharge from the intensive care unit or up to 72 hours.
  Interventions: Drug: Travesol 10%

INTERVENTIONS:
Drug: Travesol 10% — Travesol 10% (Baxter) will be administered to the post-intervention participants at a dose of 2g per kilogram of ideal body weight for up to 3 days or until the participant's discharge from the intensive care unit.
  Arms: Post-Implementation - Amino Acid Treatment

SUMMARY:
The goal of this study is to see if an infusion of amino acids given to adult male and female patients during cardiac surgery can help prevent acute kidney injury that commonly occurs when patients undergo cardiac surgery needing cardiopulmonary bypass. The main question the study aims to answer is if a short infusion of amino acids given to study participants during their scheduled heart surgery can decrease rates of acute kidney injury - which will be measured by biological markers of kidney injury in the urine.

The study will be conducted in 2 phases. Participants in the first phase will receive the current standard of anesthetic care for patients having heart surgery and markers of acute kidney injury will be measured before and after their surgery. Participants in the second group will receive the anesthetic standard of care plus a short infusion of amino acids during their surgery. They will also have markers of kidney injury measured before and after their surgery. This study is based on prior studies that showed amino acid infusions are protective against kidney injury; however, these past studies did not look at markers of kidney injury in the urine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older undergoing elective cardiac surgery requiring cardiopulmonary bypass.
* Anticipated stay of at least one night in the ICU following cardiac surgery.
* Eligible patients must have a baseline serum creatinine measurement obtained during the current hospitalization, or within 365 days of the current hospitalization.
* Patients agree to participation and completed informed consent process.

Exclusion Criteria:

* Preoperative or planned post-operative need for renal replacement therapy.
* Stage IV or greater chronic kidney disease, defined as estimated glomular filtration rate of less than 30 mL/minute per 1.73 M^2 of body surface area as calculated by the Cockcroft-Gault equation.
* Emergent cardiac surgical patients and patients undergoing orthotopic heart transplant.
* Any patient who has a history of renal transplant.
* Patients who have a documented allergy or hypersensitivity to one or more of the amino acids.
* Patients with cognitive impairment who cannot provide consent.
* Patients with congenital alteration of amino acid metabolism.
* Any patient who declines to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of acute kidney injury biomarker: tissue inhibitor of metalloproteinases 2 (TIMP-2) | In the first hour upon arrival to the ICU, following completion of surgery. On average 6 hours from start of procedure, up to 12 hours.
  Urinary TIMP-2 via NephroCheck, measured in (ng/mL)/1000.
Quantification of acute kidney injury biomarker: insulin-like growth factor-binding protein 7 (IGFBP7) | Baseline prior to cardiopulmonary bypass
  Urinary IGFBP7, measured in (ng/mL)/1000.
Quantification of acute kidney injury biomarker: insulin-like growth factor-binding protein 7 (IGFBP7) | In the first hour upon arrival to the ICU, following the completion of surgery. On average 6 hours from the start of the procedure, up to 12 hours.
  Urinary IGFBP7, measured in (ng/mL)/1000.

OTHER OUTCOMES:
Quantification of acute kidney injury biomarker: tissue inhibitor of metalloproteinases 2 (TIMP-2) | Baseline prior to cardiopulmonary bypass
  Urinary TIMP-2 via NephroCheck, measured in (ng/mL)/1000.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Adenwala, MD, Principal Investigator — Assistant Professor, Department of Anesthesiology

IPD SHARING:
Plan to Share IPD: Undecided